CLINICAL TRIAL: NCT07036237
Title: The Comparison Of The Effect Of Intracanal Rinse of Tramadol and Dexamethasone on Post-Endodontic Pain in Teeth With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Comparison Of The Effect Of Final Rinse Of Tramadol and Dexamethasone on Post-Endodontic Pain in Teeth With SIP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hassan Mirza, MDS Trainee Of Operative Dentistry, Dow University Of Health Sciences, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HMIrza
Record Dates: First submitted 2025-05-15; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Post-endodontic Pain
Keywords: Opiod analgesics; Root Canal Irrigant; Symptomatic Irreversible Pulpitis; SIP; Visual Analoque Scale; VAS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients included in the study will pick an envelope A, B or C for inclusion in the Group A, B or C. Researcher will himself be responsible for randomization and recruitment of participants into groups. In this Double blinded study neither clinician or patient will not know the drug of the envelope and the syringes will be masked by white paper labeled A, B and C by the dental assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tramadol Group (Experimental): Group A 30 participants will receive Tramadol as part of root canal treatment.
  Interventions: Drug: Dexamethasone Group
- dexamethasone group (Experimental): Dexamehasone as a final irrigant
  Interventions: Drug: Tramadol group
- Normal Saline group (Placebo Comparator): normal saline as a final irrigant
  Interventions: Drug: Tramadol group; Drug: Dexamethasone Group

INTERVENTIONS:
Drug: Tramadol group — Drug used as final irrigant
  Other Names: Drug A
  Arms: Normal Saline group; dexamethasone group
Drug: Dexamethasone Group — drug used as a final irrigant
  Other Names: Drug B
  Arms: Normal Saline group; Tramadol Group

SUMMARY:
Briefly, 105 teeth with symptomatic irreversible pulpitis will be included in the study and randomly allocated to three groups (A, B and C). Pre-Operative pain score using VAS will be taken after which root canal treatment shall be initiated. Group A (35 teeth) will receive normal saline as a final irrigant. 35 teeth each of Groups B and C will receive Dexamethasone and Tramadol Solutions, respectively as final irrigants. Post-operative pain scores will be recorded after 6, 12, 24 and 48 hours after the procedure. Statistical analysis will be performed using SPSS version 26.0. Mean comparison of pre-treatment and post-treatment VAS scores will be done by repeated measure two-way ANOVA. Post-hoc LSD test will be applied for pairwise comparison within and/or between groups.

The sample size of 105 subjects (35 including 5 as a drop out per group) is calculated using PASS version 15, based on two sample proportion with 95% confidence of interval and 80% power of test, no pain in dexamethasone (81.7%) and drug2

DETAILED DESCRIPTION:
Diagnosis of symptomatic irreversible pulpitis will be made by Clinical and radiographic examination, electric pulp test and cold test. Patients included in the study will pick an envelope A, B or C for inclusion in the Group A, B or C. Researcher will himself be responsible for randomization and recruitment of participants into groups. In this Double blinded study neither clinician or patient will not know the drug of the envelope and the syringes will be masked by white paper labeled A, B and C by the dental assistant. They will be explained briefly about the procedure, safety, usefulness of the drug and informed consent will be taken (Appendix 1 & 2 consent form). Pre-operative pain will be recorded using VAS. Treatment will be started by local anesthesia with Lidocaine 2% and Epinephrine 1:100,000 (Medicaine) and rubber dam (Medicom) isolation. Access opening will be done by EndoZ bur (Dentsply) and complete deroofing of the pulp chamber will be done.

Irrigation will be done by sodium hypochlorite 5% (i-dental) and root anal orifice will be located by DG-16 probe. #8 and #10 K-files (sybron endo) will be used for negotiating the canals. Working length will be taken by #20 K-file using apex locator(E-connect) and will be confirmed by periapical x-ray. Engine driven rotary motor (x smart, Dentsply) will be used to accomplish cleaning and shaping step of root canal treatment. Researcher will himself carry out single visit root canal treatment in mandibular teeth diagnosed symptomatic irreversible pulpitis with no peri-radicular periodontitis. Pro taper Gold (Dentsply) will be used for instrumentation with prescribed torque and rotations per minute. Root canal irrigation will be done after each step of filing with 5% sodium hypochlorite 2ml with final rinse of normal saline in all the groups. At this point, following drying the canals with paper points, Group A will receive 1ml of tramadol solution (Searle Pharma) 100mg/2ml for each canal Group B will

14

receive 1ml of dexamethasone solution (Searle Pharma) 4mg/1ml for each canal and group C will receive 1ml of normal saline solution for each canal as a final irrigant. Final irrigant will be activated with ultrasonic tip Model:E62 ENDODONTICS (Guilin Woodpecker Medical Instrument Co.Ltd) and canals will be dried with paperpoints. Filling of the canal will be done by gutta percha (Dentsply) and root canal sealer (Sealapex) by lateral compaction technique.

Permanent restoration will be placed on the same visit. Ibuprofen 400mg will be advised as a rescue oral pill and postoperative pain will be assessed by giving forms containing Visual Analogue Scale (Appendix 3) to fill at 6-, 12-,24 and 48-hours intervals. If the patient is illiterate, will be asked verbally to fill in the form. Patient will be called at the specified intervals for follow up and fill in the forms.

ELIGIBILITY:
Inclusion Criteria

* ASA 1 and ASA 2 eligible patients
* Patients aged between 18 and 50 years
* Mandibular Single rooted teeth diagnosed with symptomatic irreversible pulpitis
* Preoperative pain measured with the help of visual analogue scale and
* Only one diseased tooth within the arch Exclusion Criteria
* Patients who have taken any analgesic at least 12 hours before the procedure
* Teeth diagnosed with pulpal necrosis and periradicular periodontitis
* Teeth non restorable due to any reason,
* Root canal calcifications and resorptions.
* Women with breast feeding and pregnancy
* Patients allergic to any of the two drugs shall also be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-11-17 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Pain intensity | 6 to 48 hours
  Measurement Tool : Visual Analogue Scale (VAS) Unit Of Measure : Pain intensity will be assessed on a 0-10 scale, where 0 represents no pain and 10 represents the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad AM Amin, FCPS, Study Chair — Dow University of Health Sciences; Fazal FM Qazi, FCPS, Study Director — Dow University of Health Sciences
Locations (1):
- DIOKHS,Dow University Of Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Study will be published in a recongnized Journal to share with other researchers
Supporting Information: Study Protocol
Time Frame: 2to3years
Access Criteria: Journal